CLINICAL TRIAL: NCT02661568
Title: Anticoagulation Treatment Patterns and Persistence After Acute Venous Thromboembolism in the UK in Routine Clinical Practice: A Retrospective Database Study of the Clinical Practice Research Datalink and the Hospital Episode Statistics Dataset
Brief Title: Description of Patients With Acute Venous Thromboembolism in the UK's Clinical Practice Research Datalink Linked With Hospital Episode Statistics Dataset (CPRD-HES)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-368
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Population with condition and with exposure

SUMMARY:
This study will utilize a retrospective cohort design. Using the Clinical Practice Research Datalink (CPRD) linked with Hospital Episode Statistics (HES) datasets, all patients with a record of VTE diagnosis between 1 April, 2008 and 31 March, 2013 will be identified and followed from the occurrence of VTE (index date) to the first of 24 months after the index date, end of the study period, leaving the database, or death.

ELIGIBILITY:
Inclusion Criteria:

VTE events will be included if:

* they are identified by at least one Read code diagnosis of acute VTE in the CPRD, or one ICD-10 code of VTE in the HES database, during the study period; and
* they occurred in patients ≥ 18 years old at time of VTE occurrence; and
* CPRD acceptability quality criteria are present

Exclusion Criteria:

VTE events will be excluded if:

* Patients have fewer than 12 months of computerized data available prior to VTE occurrence. The date of start of computerized records will be the latter of the patient's date of current registration with the practice or the practice's Up-to-Standard (UTS) date (date from which practice data is of research quality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, community sample and residents of a community
Sampling Method: Non-Probability Sample
Enrollment: 38409 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Anticoagulation treatment patterns for patients following acute Venous Thromboembolism (VTE) based on all VTE events that occur during the study period | up to 24 months following VTE occurrence
  Anticoagulation treatment pattern includes type of anticoagulant (AC), duration of AC treatment, switching between ACs and switching from AC to aspirin or other antiplatelet agents (APA).

SECONDARY OUTCOMES:
Demographic characteristics (age, gender) of patients with acute VTE | up to 24 months following VTE occurrence
Clinical characteristics (comorbidities, concomitant treatments, medical and surgical history) of patients with acute VTE | up to 24 months following VTE occurrence
Rates of unplanned (emergency) hospital admission, major surgery, major bleeding, and VTE recurrence | up to 24 months following VTE occurrence
Baseline demographic and clinical characteristics associated with the duration of AC treatment after VTE | up to 24 months following VTE occurrence
Baseline demographic and clinical characteristics associated with novel oral anticoagulant (NOAC) treatment compared with vitamin K antagonist (VKA) treatment following VTE | up to 24 months following VTE occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx